CLINICAL TRIAL: NCT00293280
Title: Phase II Study of CCNU (Lomustine) in Patients With Advanced Non-Small Cell Lung Cancer and Aberrant Hypermethylation of the MGMT Gene
Brief Title: Lomustine in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: JHOC-J0336, CDR0000452787; P30CA006973 (NIH); JHOC-J0336; WIRB-20031229; WCCC-CO-00501
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; recurrent non-small cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Lomustine

INTERVENTIONS:
Drug: lomustine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as lomustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well lomustine works in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the response rate to lomustine in patients with stage IIIB or IV non-small cell lung cancer with aberrant methylation of the MGMT gene.
* Determine whether the response rate in these patients is significantly greater than that of the historical control.

Secondary

* Collect preliminary data on toxicity, disease stabilization, time to disease progression, and overall survival.

Tertiary

* Evaluate the association between clinical outcome and immunohistochemical staining by grouping the patients as complete or partial loss of MGMT gene.

OUTLINE: This is a multicenter study.

Patients receive oral lomustine once on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell bronchogenic carcinoma, including the following histologic subtypes:

  * Squamous cell
  * Adenocarcinoma
  * Adenosquamous
  * Large cell anaplastic
  * Bronchoalveolar
  * Non-small cell carcinoma not otherwise specified (NOS)
* Stage IIIB disease (with a pleural effusion) or stage IV disease

  * Stage IV patients with brain metastases are eligible provided the brain metastases are clinically stable after treatment with surgery and/or radiation therapy
* Tumors must test positive for aberrant methylation of the MGMT gene by methylation-specific polymerase chain reaction
* Bidimensionally measurable or evaluable disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* No other active malignancies
* WBC ≥ 4,000/mm^3 OR absolute neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin normal
* AST < 5 times upper limit of normal
* Serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* No uncontrolled serious active infection
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 3 weeks since prior chemotherapy
* No more than 2 prior chemotherapy regimens
* No prior therapy with nitrosoureas
* Recovered from prior radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Toxicity
Disease stabilization
Time to disease progression
Overall survival
Association between clinical outcome and immunohistochemical staining

CONTACTS AND LOCATIONS:
Overall Officials: Julie Brahmer, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States